CLINICAL TRIAL: NCT01822041
Title: 14C-ARN-509 Microdose Absolute Bioavailability and Microtracer Absorption, Metabolism, and Excretion Study in Healthy Volunteers
Brief Title: 14C-ARN-509 Microtracer Label AME and Absolute BA Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aragon Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ARN-509-006; 2012-004899-19 (EudraCT Number)
Record Dates: First submitted 2013-02-26; First posted 2013-04-02 (Estimated); Last update posted 2013-09-13 (Estimated); Status verified 2013-09

CONDITIONS: Healthy
Keywords: healthy volunteers; mass balance study; Pharmacokinetics
MeSH Terms: interventions — apalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part A - 14C labeled ARN-509 (Active Comparator): Single oral dose of 240 mg ARN-509, followed after 2 hours (at the average tmax of ARN-509) by an intravenous (i.v.) microdose of 100 μg (9.25 kBq, 250 nCi) 14C-ARN-509
  Interventions: Drug: ARN-509
- Part B: 14C labeled ARN-509 (Active Comparator): Single oral dose of 240 mg ARN-509, followed after 2 hours (at the average tmax of ARN-509) by an oral dose of 240 mg ARN-509 with 37 kBq (1000 nCi) of 14C-ARN-509
  Interventions: Drug: ARN-509

INTERVENTIONS:
Drug: ARN-509 — Single oral dose of 240 mg ARN-509

SUMMARY:
This is study in healthy human volunteers to determine the absorption, metabolism, and excretion (AME) profile of ARN-509 as well as its absolute oral bioavailability (BA).

DETAILED DESCRIPTION:
Two cohorts of 6 healthy volunteers will be enrolled for the AME and absolute BA parts, respectively. The dose for both cohorts is 240 mg. The expected exposure of the dose is 7-fold lower than the steady state reached in patients with castration-resistant prostate cancer.

ELIGIBILITY:
Key Inclusion Criteria:

1. Gender : male
2. Age : 50 - 80 years, inclusive
3. Body Mass Index (BMI) : 18.5-30.0 kg/m2
4. Ability and willingness to abstain from alcohol, methylxanthine-containing beverages or food (coffee, tea, cola, chocolate, "power drinks"), grapefruit (juice) and tobacco products from 48 h prior to entry in the clinical research center until discharge
5. Medical history without major pathology

Key Exclusion Criteria:

1. Evidence of clinically relevant pathology.
2. Mental handicap.
3. History of relevant drug and/or food allergies.
4. Regular/routine treatment with non-topical medications within 30 days prior to entry into the clinical research center.
5. Smoking.
6. History of alcohol abuse or drug addiction (including soft drugs like cannabis products).
7. Use of concomitant medication, except for acetaminophen (paracetamol) and topical medications
8. Irregular defecation pattern (less than once per 2 days).
9. Positive drug screen (opiates, methadone, cocaine, amphetamines, cannabinoids, barbiturates, benzodiazepines, and alcohol).
10. Intake of more than 24 units of alcohol per week (one unit of alcohol equals approximately 250 mL of beer, 100 mL of wine or 35 mL of spirits).
11. Positive screen on HBsAg, anti-HCV or anti-HIV 1/2.
12. Illness within five days prior to drug administration.

Ages: 50 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-03; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Mass Balance | 2 months 10 days
  To determine the rate and routes of excretion of ARN-509 in urine, feces, and expired air
Absolute Oral Bioavailability | 2 months 10 days
  To determine absolute oral bioavailability of ARN-509

SECONDARY OUTCOMES:
Metabolite Profile | 2 months 10 days
  To identify and quantify the ARN-509 metabolites in plasma, urine, and feces

CONTACTS AND LOCATIONS:
Overall Officials: Nada al Kotbi, MD, Principal Investigator — PRA International Group BV; Helen Pruim-Tait, MA, MSc, Study Director — PRA International Group BV
Locations (1):
- PRA - Clinical Research Unit, University Medical Centre Groningen, Groningen, Netherlands